CLINICAL TRIAL: NCT01096225
Title: Study of Humoral and Cellular Immunogenicity of Split-vaccine to Swine-origin H1N1 Influenza
Brief Title: Immunogenicity Study of S-OIV H1N1 Influenza Vaccine
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Hualan Biological Bacterin Co. Ltd. (Industry); Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Institute of Microbiology, Chinese Academy of Sciences
Other Study IDs: Immunity_S-OIV_A/H1N1_vaccine
Record Dates: First submitted 2010-03-29; First posted 2010-03-31 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-03

CONDITIONS: Human Influenza
Keywords: the antibody response; T-cell response; S-OIV; vaccine; Immunogenicity assessment
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Peripheral Blood Mononuclear Cell (PBMC)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- vaccinated group
  Interventions: Biological: split-virion, H1N1 vaccine of 15 μg

INTERVENTIONS:
Biological: split-virion, H1N1 vaccine of 15 μg — split-virion inactivated S-OIV vaccine of 15 μg on day 0 and 21.
  Other Names: S-OIV vaccine

SUMMARY:
The primary immunogenicity objective is to assess the antibody response and T-cell response of split-virion inactivated A (H1N1) vaccine. Participants will include up to 20 healthy persons of age 20 and older who have no history of novel influenza H1N1 2009 infection in latest 3 months or novel influenza H1N1 2009 vaccination. This is a randomized study in healthy males and non-pregnant females, aged 20 years and older. All subjects will be stratified into 1 dose group (15mcg per dose), and will receive intramuscular influenza H1N1 vaccine. The H1N1 vaccine will be administered at Day 0 and Day 21. On Day 0, Day 10, Day 21, Day 28, Day 35 and Day 42 after first vaccination (Day 0), the immunogenicity testing will be manipulated. The antibody response of immunogenicity testing will be hemagglutination inhibiting (HAI) on serum. The T-cell response will be interferon-gamma ELISPOT assay and Tetramer staining using PBMCs.

DETAILED DESCRIPTION:
In 2009, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in North America. It rapidly spread to many countries around the world, which soon meets the World Health Organization (WHO) criteria for a pandemic. Data from several clinical trails with the split-virion inactivated S-OIV vaccine suggest that the vaccine stimulated strong specific antibody against S-OIV. However, the is no T-cell response data after the vaccination. In addition, we do not know S-OIV specific cellular immunity level of the population. These facts indicate the need to assess both the antibody response and T-cell response after the vaccination of the split-virion inactivated S-OIV vaccine. The primary immunogenicity objective is to assess the antibody response and T-cell response of split-virion inactivated A (H1N1) vaccine. Participants will contain only one age group, including up to 20 healthy persons of age 20 and older who have no history of novel influenza H1N1 2009 infection in latest 3 months or novel influenza H1N1 2009 vaccination. This is a randomized study in healthy males and non-pregnant females. All subjects will be stratified into 1 dose group (15mcg per dose), and will receive intramuscular influenza H1N1 vaccine. The H1N1 vaccine will be administered at Day 0 and Day 21. On Day 0, Day 10, Day 21, Day 28, Day 35 and Day 42 after first vaccination (Day 0), the immunogenicity testing will be manipulated. The antibody response of immunogenicity testing will be hemagglutination inhibiting (HAI) on serum. The T-cell response will be interferon-gamma ELISPOT assay and Tetramer staining using PBMCs.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female aged 20 and older
2. Be able to show legal identity card for the sake of recruitment
3. Volunteers or their guardians are able to understand and sign the informed consent

Exclusion Criteria:

1. Cases, cured cases and close contact of influenza A (H1N1) virus
2. Women of pregnancy, lactation or about to be pregnant in 60 days
3. Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, such as egg, egg protein, etc
4. Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
5. Autoimmune disease or immunodeficiency
6. Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
7. Diabetes mellitus (type I or II), with the exception of gestational diabetes
8. History of thyroidectomy or thyroid disease that required medication within the past 12 months
9. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years
10. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
11. Active malignancy or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of study
12. Seizure disorder other than:

    * Febrile seizures under the age of two years old
    * Seizures secondary to alcohol withdrawal more than 3 years ago, or
    * A singular seizure not requiring treatment within the last 3 years
13. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
14. Guillain-Barre Syndrome
15. Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
16. History of any blood products or swine-origin H1N1 or seasonal influenza vaccine administration within 3 months before the dosing
17. Administration of any other investigational research agents within 30 days before the dosing
18. Administration of any live attenuated vaccine within 30 days before the dosing
19. Administration of subunit or inactivated vaccines, e.g., pneumococcal vaccine, or allergy treatment with antigen injections, within 14 days before the dosing
20. Be receiving anti-TB prophylaxis or therapy currently
21. Axillary temperature > 37.0 centigrade at the time of dosing
22. Psychiatric condition that precludes compliance with the protocol:

    * Past or present psychoses
    * Past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years
    * Disorder requiring lithium
    * Suicidal ideation occurring within five years prior to enrollment
23. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Volunteers of age 20 and older who have no history of novel influenza H1N1 2009 infection in latest 3 months or novel influenza H1N1 2009 vaccination.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-04 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Assess the immunity level of the subjects before vaccination. | On Day 0 after first vaccination
  hemagglutination inhibiting (HAI), ELISPOT and Tetramer staining.

SECONDARY OUTCOMES:
Assess the immunity level of the subjects 10 days after vaccination | On Day 10 after first vaccination
  hemagglutination inhibiting (HAI), ELISPOT and Tetramer staining.
Assess the immunity level of the subjects 21 days after vaccination | On Day 21 after first vaccination
  hemagglutination inhibiting (HAI), ELISPOT and Tetramer staining.
Assess the immunity level of the subjects 28 days after vaccination | On Day 28 after first vaccination
  hemagglutination inhibiting (HAI), ELISPOT and Tetramer staining.
Assess the immunity level of the subjects 35 days after vaccination | On Day 35 after first vaccination
  hemagglutination inhibiting (HAI), ELISPOT and Tetramer staining.
Assess the immunity level of the subjects 42 days after vaccination | On Day 42 after first vaccination
  hemagglutination inhibiting (HAI), ELISPOT and Tetramer staining.

CONTACTS AND LOCATIONS:
Overall Officials: George Fu Gao, Ph.D., Principal Investigator — CAS Key Laboratory of Pathogenic Microbiology and Immunology,Institute of microbiology, Chinese Academy of Sciences
Locations (1):
- Institute of microbiology, Chinese Academy of Sciences, Beijing, Beijing Municipality, China